CLINICAL TRIAL: NCT04974255
Title: Does Gluten Sensitivity Play a Role in Development of Thyroiditis
Brief Title: Association of TTGA (Tissue Transglutaminase Antibody) and Histopathologic Findings in Thyroidectomy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gorkem Gundogan, MD, Senior Resident of General Surgery, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 59/02
Record Dates: First submitted 2021-05-31; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Thyroid Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Operated Patients (Experimental): Measurement of fibrosis degree and Anti-tTG levels
  Interventions: Other: Measuring of fibrosis in thyroid specimen and measuring of Anti-tTG in serum samples

INTERVENTIONS:
Other: Measuring of fibrosis in thyroid specimen and measuring of Anti-tTG in serum samples — Examination of pathology specimen and laboratory measuring

SUMMARY:
Gluten sensitivity is the most common auto-immune disease associated with auto-immune thyroiditis. This association is through elevated anti-Tissue transglutaminase (Anti-tTG) levels both in Celiac disease and thyroiditis. In our study we tried to find if there is any correlation in between Anti-tTG and degree of fibrosis in thyroid tissue (Post-operative specimen).

DETAILED DESCRIPTION:
Most common auto-immune disease associated with Celiac disease is autoimmune thyroiditis. This association in between Celiac disease and aout-immune thyroiditis is related with asymptomatic rise in anti-tTG levels. In our study, we planned to show that if there is any correlation of thyroiditis related fibrosis in thyroid tissue with anti-tTG IgA ( immune-globulin A) and IgG (immune-globulin G).

ELIGIBILITY:
Inclusion Criteria:

* Thyroiditis patients operated for any indication

Exclusion Criteria:

* Patients with known IgA deficiency

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-07-26 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Amount of fibrosis in thyroid tissue and measured level of anti-tTG levels in serum | one day after operation
  Degree of fibrosis was defined after painting of slides with masson trichrome as absent, mild, moderate semi-quantitatively.
Measurement of Anti-tTG levels in serum | one day after operation
  Amount of serum Anti-TG in IU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Gorkem Gundogan, Principal Investigator — Not Affliated
Locations (1):
- SBU Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Hospital records
Supporting Information: SAP, ICF, CSR
Time Frame: June 2021 for 1 year
Access Criteria: No criteria